CLINICAL TRIAL: NCT02741232
Title: Comparison of Perioperative Opioid Consumption Following Pectoral Nerve Block Under General Anesthesia for Breast Cancer Surgery: A Randomized Clinical Trial
Brief Title: Comparison of Perioperative Opioid Consumption Following Pectoral Nerve Block for Breast Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, Olivier Verdonck, Clinical Assistant Professor, Maisonneuve-Rosemont Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15075
Record Dates: First submitted 2016-04-13; First posted 2016-04-18 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Nerve Block; Mastectomy
Keywords: analgesics, opioids; pectoral block
MeSH Terms: interventions — Lidocaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pectoral nerve block (Active Comparator): After induction of general anesthesia and under ultrasound visual guidance, pectoral block is performed with 30 mL total of local anesthetic (1% lidocaine + 1/400000 epinephrine). 10 mL of local anesthetic between pectoralis major muscle and pectoralis minor muscle and 20 mL between pectoralis minor muscle and serratus anterior muscle at the third rib.
  Interventions: Drug: Lidocaine 1% with epinephrine 1/400000
- Sham block (Sham Comparator): No needle or injection will be used
  Interventions: Other: sham block

INTERVENTIONS:
Drug: Lidocaine 1% with epinephrine 1/400000
  Other Names: xylocaine with epinephrine
  Arms: Pectoral nerve block
Other: sham block
  Arms: Sham block

SUMMARY:
In this study, the investigators will compare the intraoperative opioid consumption for patients undergoing breast cancer surgery. The patients will be divided in two groups, the first one will receive a pectoral nerve block right after induction of anesthesia and the second one, the control group, will not receive the pectoral block. Our hypothesis is that the pectoral nerve block reduces the opioid consumption during the surgery.

DETAILED DESCRIPTION:
After induction of general anesthesia with propofol, remifentanil and succinylcholine, the patients will be divided either in the pectoral block group or the control group (sham block). Both groups will receive the same perioperative and postoperative anesthetic protocol. The investigator in charge of the patient will leave the operative room right before the completion of the pectoral block (or the sham block) to preserve randomisation and the block will be performed by another investigator. The pectoral block is performed under ultrasound guidance with 10 cc of lidocaine 1% with epinephrine 1/400000 between the pectoralis major muscle and the pectoralis minor muscle and 20 cc of the same solution between the pectoralis minor muscle and the serratus anterior muscle at the third rib. Anesthesia will be maintained with sevoflurane for a bispectral (BIS) index between 45 and 60. Analgesia will be provided with a perfusion of remifentanil adjusted to maintain a mean arterial blood pressure (MAP) in the range of ± 10% of the basal MAP (mean of the last three MAPs obtained before surgical incision, under sevoflurane-only anesthesia). The total remifentanil consumption will be assessed and compared between the groups. The investigators believe that the pectoral nerve block will significantly reduce the intraoperative remifentanil consumption.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 to 3 inclusively
* breast cancer surgery with or without axillary dissection

Exclusion Criteria:

* any contraindication to the pectoral nerve block (coagulopathy, infection, pre- existing neuropathy, local anesthetic allergy and refusal of local anesthesia)
* refusal to participate in the study
* patient with dementia
* preoperative breast pain
* preoperative opioid consumption
* breast reconstructive surgery
* bilateral surgery
* pregnant patient

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-03; Primary Completion 2017-08-30 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
Intraoperative remifentanil consumption for the first 30 minutes of surgery | 30 minutes

SECONDARY OUTCOMES:
Total intraoperative remifentanil consumption | 2 hours
Total intraoperative sevoflurane consumption | 2 hours
Postoperative pain evaluation | 30 minutes
  using the numerical rating scale
Postoperative nausea and vomiting evaluation | 30 minutes
Total time in the recovery room | 60 minutes
Postoperative opioid consumption | 1 hour
  dilaudid consumption

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Maisonneuve-Rosemont, Montreal, Quebec, Canada